CLINICAL TRIAL: NCT07356336
Title: Examining the Efficacy of a Personalized Cognitive Model as Non-Pharmacological Intervention for Behavioral and Psychological Symptoms of Dementia
Brief Title: Cognitive Model for Behavioral Interventions as a Non-pharmacological Intervention for Behavioral and Psychological Symptoms of Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Alexianen Zorggroep Tienen (Unknown); vzw Bejaardenzorg Grauwzusters Limburg (Unknown); Mondriaan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25398_CoMBI_BPSD_WZC
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Behavioral and Psychological Symptoms of Dementia
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention): Participants receive standard care without implementation of a theory-based, behavioral counseling intervention.
- CoMBI (Experimental)
  Interventions: Behavioral: CoMBI

INTERVENTIONS:
Behavioral: CoMBI — CoMBI describes a four-step approach. First, the primary caregiver systematically observes and assesses the resident's BPSD using the NPI-Q. Second, the person's core needs are identified. An informant completes the PID-5-BF+M. The results of the PID-5-BF+M together with the overview of the different personality types, help identify the resident's core needs. Third, the care team selects one core need based on the most prominent and challenging BPSD. They choose a maximum of three interventions, which can focus on the substantive contact, attitude and environment of the resident. Finally, The selected interventions are further specified and personalized so that they are appropriate for the person with dementia, taking into account their life history This is documented in a CoMBI care plan, specifying which interventions will be applied and the desired behavioral outcomes.
  Arms: CoMBI

SUMMARY:
The goal of this study is to evaluate whether the Cognitive Model for Behavioral Interventions (CoMBI), a person-centered, non-pharmacological intervention, can reduce behavioral and psychological symptoms of dementia (BPSD) in people with dementia living in nursing homes. The study also aims to examine whether CoMBI can reduce caregiver burden and improve quality of life in people with dementia.

The main questions it aims to answer are:

Does CoMBI reduce the severity of behavioral and psychological symptoms of dementia compared to care as usual?

Does a reduction in BPSD lead to lower caregiver burden and improved quality of life for people with dementia?

Do personal factors, such as personality (dys)functioning, gender, level of cognitive impairment and stage of dementia, influence the effectiveness of CoMBI?

Researchers will compare CoMBI to care as usual to determine whether CoMBI leads to better outcomes for people with dementia and their caregivers.

Participants will:

Receive care in residential long-term care facilities where care staff are trained to apply CoMBI.

Be observed and assessed repeatedly over time as part of a stepped-wedge cluster randomized trial design.

DETAILED DESCRIPTION:
Behavioral and Psychological Symptoms of Dementia (BPSD), also referred to as neuropsychiatric symptoms, are highly prevalent across all types of dementia and represent a major clinical and societal challenge. These symptoms are associated with accelerated disease progression, reduced quality of life for people with dementia, and substantial burden for both formal and informal caregivers. In residential long-term care facilities, where BPSD are particularly common, management often relies heavily on psychotropic medication despite risks, including increased morbidity and mortality. International guidelines therefore recommend person-centered, non-pharmacological interventions as first-line treatment. However, existing non-pharmacological approaches show mixed effects, face implementation barriers, and often insufficiently account for individual differences such as premorbid personality, despite growing evidence that personality plays a key role in the development and severity of BPSD.

The Cognitive Model for Behavioral Interventions (CoMBI) is a person-centered, non-pharmacological intervention designed to address these limitations. CoMBI is grounded in the assumption that BPSD partly emerge when underlying core needs are insufficiently met. These core needs are shaped by premorbid personality characteristics and are activated by specific environmental triggers. Drawing on Beck's cognitive model of personality disorders and nursing interventions from the Nursing Intervention Classification, CoMBI distinguishes distinct personality profiles, each associated with characteristic unmet needs and triggering situations. For each profile, tailored intervention strategies have been developed to compensate for unmet needs by modifying environmental factors and caregiver responses.

The CoMBI training provides caregivers with a structured framework to understand BPSD in relation to premorbid personality and unmet core needs. Care staff are trained to assess BPSD, identify personality-related core needs and triggering events, and implement tailored interventions. This is well documented in a CoMBI care plan, specifying which interventions will be applied and the desired behavioral outcomes. The care plan can be reevaluated every care team meeting.

To empirically demonstrate the effectiveness of CoMBI, we will conduct a stepped-wedge cluster randomized trial (SW-CRT) with repeated measures. All units of the participating nursing homes will initially receive care as usual (CAU) and will sequentially transition to the CoMBI condition. Outcome measurements will be conducted every four weeks, including at the time each unit changes from CAU to CoMBI. Outcomes are assessed using the Neuropsychiatric Inventory Questionnaire (NPI-Q), the Global Deterioration Scale (GDS), Qualidem and the Montreal Cognitive Assessment (MoCA). To properly identify the core needs for CoMBI, two personality questionnaires will be administered, namely the Personality Inventory for DSM-5 Brief Form + Modified (PID-5-BF+M) and the Level of Personality Functioning Scale Brief Form 2.0 (LPFS-BF 2.0).

ELIGIBILITY:
Inclusion Criteria:

* Being a resident in a participating nursing home
* Having a formal diagnosis of neurocognitive disorder (NCD) accord-ing to DSM-5-TR (e.g. Alzheimer's disease, NCD with Lewy Bodies, Vascular NCD, …) or a medical record indicating probable dementia
* Presence of one or more BPSD symptoms at moment of inclusion in the study (measured with the NPI-Q at baseline). Symptoms measured by the NPI-Q include delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria/elated mood, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, nighttime behavior disturbances/sleep disturbances, and changes in appetite and eating behavior.
* Primary caregivers (i.e. nurses providing daily care) and patient's representative and/or a close relative/friend (i.e. informant who will fill in the premorbid personality questionnaire) are proficient in Dutch (i.e., are able to fill in the questionnaires)
* The informant who fills in the premorbid personality questionnaire knows the patient well from before the onset of neurocognitive problems
* As individuals with dementia are often legally incapacitated, informed consent will be obtained prior to participation from the resident when competent to consent, or otherwise from the resident's legal representative when legally incompetent.

Exclusion Criteria:

Exclusion criterion for nursing homes is:

- Already applying a structured (theory-based) behavioral counseling as CAU.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory - Questionnaire (NPI-Q) | Before the start of CAU, before the start of CoMBI and after four weeks of CoMBI training.
  The Neuropsychiatric Inventory - Questionnaire (NPI-Q) (de Jonghe et al., 2003; Kaufer et al., 2000) is a validated informant evaluation of BPSD measuring severity (rating 0-3) and caregiver distress (0-5) of 12 BPSD domains (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturb-ance, nighttime behaviors, appetite/eating).
Qualidem | Before the start of CAU, before the start of CoMBI and after four weeks of CoMBI training.
  The Qualidem (Ettema et al., 2007) is a forty-item validated behavior observation-scale for patients (i.e. nursing homes) with up to severe dementia and can be administered in 15 minutes. Nine sub-scales (care relationship, positive affect, negative affect, restless tense behavior, positive self-image, social relations, social isolation, feeling at home, having something to do) provide a QoL-profile that can be used to evaluate the effects of intervention.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Before the start of CAU, before the start of CoMBI and after four weeks of CoMBI training.
  The MoCA is a brief (10-15 minute) 30-point cognitive screening instrument which has been prov-en useful in identifying cognitive symptoms associated with dementia.
the Global Deterioration Scale | Before the start of CAU, before the start of CoMBI and after four weeks of CoMBI training.
  The GDS, describes clinical characteristics (e.g., memory, sleep, social impairment) for stages of cognitive function for those suffering from a primary degenerative dementia. Primary caregivers estimate the level of where an individual is in the disease process by observing that individual's behavioral characteristics and comparing them to the GDS stage descriptions.
the Level of Personality Functioning-scale brief form 2.0 informant version (LPFS-BF 2.0) | Before the start of CAU, before the start of CoMBI and after four weeks of CoMBI training.
  Higher total scores indicate higher dysfunctioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexianen Zorggroep Tienen, Tienen, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No